CLINICAL TRIAL: NCT06793995
Title: A Phase 1 Study to Evaluate the Effect of Food and Age on the Pharmacokinetics of LPM526000133 Fumarate Capsules (LY03017) in Healthy Volunteers
Brief Title: Effect of Food and Age on the Pharmacokinetics of LY03017
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LY03017/CT-CHN-102
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer's Disease Psychosis; Parkinson Disease Psychosis; Negative Symptoms of Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LY03017 (Part A, fasting-fed) (Experimental): Subjects will be administrated 40 mg of LY03017 under fasting conditions and fed conditions in period 1 and 2 respectively. There will be a 7-day washout period between the first and second dose.
  Interventions: Drug: LY03017
- LY03017 (Part A, fed-fasting) (Experimental): Subjects will be administrated 40 mg of LY03017 under fed conditions and fasting conditions in period 1 and 2 respectively. There will be a 7-day washout period between the first and second dose.
  Interventions: Drug: LY03017
- LY03017 (Part B) (Experimental): Subjects will be administrated 40 mg of LY03017 under fasting conditions on Day 1.
  Interventions: Drug: LY03017

INTERVENTIONS:
Drug: LY03017 — single dose，administered orally for each period
  Arms: LY03017 (Part A, fasting-fed); LY03017 (Part A, fed-fasting)
Drug: LY03017 — single dose，administered orally
  Arms: LY03017 (Part B)

SUMMARY:
This study consists of 2 parts. Part A is a randomized, open-label, 2-period, crossover study to evaluate the food effect of LY03017 in healthy adults. Part B is a single-arm study to evaluate the safety and pharmacokinetics of LY03017 in elderly volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject who voluntarily participate and sign the informed consent form.
* Part A：Age ≥18 and ≤ 45 years, male and female.
* Part B：Age ≥65 years, male and female.
* Body weight ≥ 50.0 kg for men and ≥ 45.0 kg for women, and body mass index (BMI) ≥18.5 and < 28.0 kg/m2.
* Able to comply with the lifestyle restrictions.

Exclusion Criteria:

* Subject has a history of allergy to any component of the investigational drug or similar drugs, or allergic constitution.
* Part A：Subject has a history of clinically significant medical conditions that may interfere with the study results, including but not limited to blood system, circulatory system, digestive system, urinary system, respiratory system, nervous system, immune system, endocrine system, malignant tumors, mental disorders and metabolic disorders.
* Part B：Subject has a history of clinically significant medical conditions that may interfere with the study results, including but not limited to blood system, circulatory system, digestive system, urinary system, respiratory system, nervous system, immune system, endocrine system, malignant tumors, mental disorders and metabolic disorders. Subjects with well-controlled, chronic and stable medical conditions (e.g., hypertension, type 2 diabetes, hyperlipidaemia) which are not expected to compromise subject safety or interfere with the study results will not be excluded.
* Any surgical condition or condition may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects.
* Subject has clinically significant abnormalities in vital signs, laboratory tests, and ECGs, such as

  1. Pulse < 55 beats/min or > 100 beats/min,
  2. Systolic blood pressure < 90 mmHg or ≥140 mmHg, Diastolic blood pressure < 60 mmHg or ≥90 mmHg,
  3. QT interval (QTc) ≥450 ms.
  4. Part B：aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or total bilirubin > 1.5 × upper limit normal (ULN), or estimated glomerular filtration rate（eGFR） <60 mL/min/1.73 m2
* Part A：Subject has used any of over-the-counter products within 7 days or prescription medications within 28 days prior to dosing.
* Part B：Subject has used any of over-the-counter products within 7 days or prescription medications within 28 days prior to dosing, with the exception of concomitant drugs for the well-controlled, chronic and stable medical conditions.
* Subject has a history of surgery within 3 months prior to administration, or failure to recover from surgery, or having an expected surgical plan during the trial.
* Subject positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab), or syphilis seroreactivity (Trust).
* Subject has a history of alcohol abuse within 1 year or positive alcohol breath test results.
* Subject has a history of substance abuse within 1 year or a positive urine drug screen.
* Subject who has daily smoking of ≥ 5 cigarettes within 3 months.
* Subject who has special requirements for food, cannot comply with the unified diet or have dysphagia.
* Subject who has consumption of special diet (such as grapefruit, chocolate, coffee, xanthine-rich foods/drinks) within 48 hours prior to dosing and/or subject who has excessive daily consumption of tea, coffee, grapefruit juice, caffeinated beverages for nearly 3 months.
* Subject who has participated in other clinical trials within 3 months before administration.
* Subject has used blood products or being blood donor or blood loss within 3 months.
* Pregnant, lactating women, or positive pregnancy test.
* Subject who refusal to contraception, or plan to donate sperm or ovums.
* Subject who has a history of needle or blood faintness.
* Subject directly involved in this clinical trial.
* Poor compliance or other conditions which would make participation in the study unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of LPM526000133 in plasma | Up to 96 hours after the last dose
The area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of LPM526000133 in plasma | Up to 96 hours after the last dose
Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC[0-last]) of LPM526000133 in plasma | Up to 96 hours after the last dose

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Up to 96 hours after the last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China